CLINICAL TRIAL: NCT05216549
Title: Water and Land-based Exercise for Children With Post COVID-19 Condition
Acronym: postcovidkids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Józef Piłsudski University of Physical Education (Other)
Collaborators: Polish National Agency for Academic Exchange (Unknown); University of Sydney (Other)
Responsible Party: Principal Investigator, Anna Ogonowska-Słodownik, Principal Investigator, Józef Piłsudski University of Physical Education
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BPN/GIN/2021/1/00071/U/00001
Record Dates: First submitted 2022-01-26; First posted 2022-01-31 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: COVID-19; Children, Only; Lung Function Decreased; Quality of Life
MeSH Terms: conditions — COVID-19; Respiratory Insufficiency

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Water-based exercise (Experimental): The water-based exercise group will be held twice a week, 45 min per session for 8 weeks. Supervised exercise will be led by the experienced physiotherapist and water-based exercise by physiotherapist with aquatic exercise expertise.Each session will consist of warm up (10 min), main part (30 min) and cool-down (5 min). During warm up children will perform lower and upper limbs aerobics and breathing exercises. The main part will consist of endurance exercises of upper and lower limbs with focus on breathing pattern. During cool-down focus will be on upper limb and thoracic cage stretches and breathing control.
  Interventions: Other: Water-based exercise
- Land-based exercise (Experimental): The land-based exercise group will be held twice a week, 45 min per session for 8 weeks. Supervised exercise will be led by the experienced physiotherapist and water-based exercise by physiotherapist with aquatic exercise expertise.Each session will consist of warm up (10 min), main part (30 min) and cool-down (5 min). During warm up children will perform lower and upper limbs aerobics and breathing exercises. The main part will consist of endurance exercises of upper and lower limbs with focus on breathing pattern. During cool-down focus will be on upper limb and thoracic cage stretches and breathing control.
  Interventions: Other: Land-based exercise
- Control (No Intervention): The control group will be asked not to change their physical activity for 8 weeks. After that period and post-test the control group will receive the exercise.

INTERVENTIONS:
Other: Water-based exercise — 8 weeks x 2 times per week for 45 min
  Arms: Water-based exercise
Other: Land-based exercise — 8 weeks x 2 times per week for 45 min
  Arms: Land-based exercise

SUMMARY:
The latest data indicate that post COVID-19 condition is frequent in children and adolescents, with the most common symptoms being fatigue, shortness of breath, exercise intolerance and weakness. Evidence that COVID-19 can have significant long-term effects on children's health highlights the need for measures to reduce the impact of the pandemic on children, ensuring that they receive appropriate treatments. Those experiencing post COVID-19 condition require more tailored exercise-related advice and improved support to be able to resume activities important to their individual well-being. To the best of our knowledge, no studies have yet addressed the issue of exercise programs for children with post COVID-19 condition.

The aim of this study, therefore, is to evaluate the effectiveness of different interventions on pulmonary function, exercise capacity, fatigue and quality of life in children with post COVID-19 condition.

This will be a randomized controlled study with pre and post intervention assessment. Children will be recruited from primary schools and primary health care units in Warsaw. Participants meeting the inclusion criteria will be randomized to one of 3 groups: water-based exercise, land-based exercise or control (no exercise). The water-based and land-based exercise groups will be held twice a week, 45 min per session for 8 weeks. Participants will be assessed at baseline and immediately post-intervention in terms of changes in pulmonary function, exercise capacity, fatigue and quality of life. Research outcomes will build the evidence-based practice for health professionals.

ELIGIBILITY:
Inclusion Criteria:

* presenting symptoms of post-COVID-19 condition confirmed by the diagnosis by general practitioner (including obligatory fatigue and shortness of breath/respiratory problems)
* age 10-12 yrs old
* adapted to aquatic setting
* <12 pts in the Ruffier test

Exclusion Criteria:

* contraindications to exercise
* chest pain
* physical activity trainings more than 2 times per week one month prior the study

Ages: 10 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 75 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-06-05 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Exercise capacity | 8 weeks (post intervention)
  Exercise capacity will be measured with the use of modification of the Balke treadmill protocol previously validated on a large population-based sample of children ages 7-18 years. Breathing parameters will be measured continuously by the "breath-to breath" method using an ergospirometer Cortex MetaMax 3B system (Biophysik GmbH, Leipzig, Germany). Output from the gas analyses will be sampled at 15 s intervals and stored for use in the calculation of the Oxygen-Uptake Efficiency Slope (OUES).
Fatigue | 8 weeks (post intervention)
  The fatigue will be assessed with the Polish adaptation of the Chronic Fatigue Syndrome Questionnaire. The questionnaire allows to determine the level of chronic fatigue and severity of individual symptoms: general fatigue, decreased vitality, mental overload, somatic symptoms, anxiety and discouragement. It includes 59 statements with one of the possible answers: "never", "sometimes", "often" - the answers are assigned the values 0, 1, 2, respectively. The higher the score, the greater the severity of the symptoms of chronic fatigue.

SECONDARY OUTCOMES:
Health-related quality of life | 8 weeks (post intervention)
  Health-related quality of life will be assessed with the PedsQL - a brief, standardized, generic assessment instrument that systematically assesses perception of HRQOL in healthy children and adolescents and those with acute and chronic health conditions.
Forced vital capacity (FVC) | 8 weeks (post intervention)
  FVC will be measured using the MES Lung Handy spirometer. Measurements will be repeated three times at five-minute intervals, and the highest score will be selected for analysis.
Forced expiratory volume/one second (FEV 1) | 8 weeks (post intervention)
  FEV 1 will be measured using the MES Lung Handy spirometer. Measurements will be repeated three times at five-minute intervals, and the highest score will be selected for analysis.
Maximal expiratory flow at 25% of forced vital capacity (MEF25) | 8 weeks (post intervention)
  MEF25 will be measured using the MES Lung Handy spirometer. Measurements will be repeated three times at five-minute intervals, and the highest score will be selected for analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Ogonowska-Slodownik, PhD, Principal Investigator — Józef Piłsudski University of Physical Education in Warsaw
Locations (1):
- Jozef Pilsudski University of Physical Education in Warsaw, Warsaw, Poland

REFERENCES:
- [Result] Ogonowska-Slodownik A, Labecka MK, Kaczmarczyk K, McNamara RJ, Starczewski M, Gajewski J, Maciejewska-Skrendo A, Morgulec-Adamowicz N. Water-Based and Land-Based Exercise for Children with Post-COVID-19 Condition (postCOVIDkids)-Protocol for a Randomized Controlled Trial. Int J Environ Res Public Health. 2022 Nov 4;19(21):14476. doi: 10.3390/ijerph192114476. PMID 36361362